CLINICAL TRIAL: NCT02804399
Title: A Phase One, Open Label, Two-period, Two-treatment, Fixed Sequence, Cross-over Study To Estimate The Effect Of Multiple Dose Rifampin On The Single Dose Pharmacokinetics Of Pf-06463922 In Healthy Volunteers.
Brief Title: A Study To Evaluate The Effect Of Rifampin On Pharmacokinetics Of PF-06463922 In Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: B7461011; RIFAMPIN DDI STUDY (Other: Alias Study Number)
Record Dates: First submitted 2016-06-10; First posted 2016-06-17 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2019-01-25 (Actual); Status verified 2018-08

CONDITIONS: Healthy
Keywords: rifampin; pharmacokinetics; PF-06463922; drug interaction
MeSH Terms: interventions — lorlatinib; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- all subjects (Experimental): subjects will receive a 100 mg single oral dose of PF-06463922 followed by a 100 mg single dose of PF-06463922 combined with 600 mg QD dose of rifampin with at least 10 days of washout period between two PF-06463922 doses.
  Interventions: Drug: PF-06463922; Drug: rifampin

INTERVENTIONS:
Drug: PF-06463922 — 100 mg oral dose on day 1 in period 1 and on day 8 in period 2
  Other Names: lorlatinib
Drug: rifampin — 600 mg QD from day 1 to day 12 in period 2.
  Other Names: rifampicin

SUMMARY:
The purpose of this study is to estimate the effect of rifampin on the single dose PK of PF-06463922.

DETAILED DESCRIPTION:
This will be a Phase 1, open-label, 2-period, 2-treatment, fixed-sequence, cross-over study in approximately 12 healthy subjects employing administration of a single oral dose of PF-06463922 in the fasted state alone, and with multiple dosing of rifampin 600 mg once a day to estimate the effect of multiple dose rifampin on the single dose PK of PF-06463922.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects of non-childbearing potential and/or male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lbs)

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease
* Any condition possibly affecting drug absorption
* Positive urine drug screen
* History of HIV, Hep B or Hep C
* History of regular alcohol consumption
* History of cardiac arrhythmia, history of AV block, history of symptomatic bradycardia, history of QTc prolongation
* History of pancreatitis or hyperlipidemia, elevated lipase

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer New Haven Clinical Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Chen J, Xu H, Pawlak S, James LP, Peltz G, Lee K, Ginman K, Bergeron M, Pithavala YK. The Effect of Rifampin on the Pharmacokinetics and Safety of Lorlatinib: Results of a Phase One, Open-Label, Crossover Study in Healthy Participants. Adv Ther. 2020 Feb;37(2):745-758. doi: 10.1007/s12325-019-01198-9. Epub 2019 Dec 20. PMID 31863284
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B7461011&StudyName=A+Phase+One%2C+Open+Label%2C+Two-period%2C+Two-treatment%2C+Fixed+Sequence%2C+Cross-over+Study+To+Estimate+The+Effect+Of+Multiple+Dose+Rifampin+On+The+Single+Dose+Pharmacokinetics+Of+Pf-06463922+In+Healthy+Volunteers.

RESULTS

PARTICIPANT FLOW:
Groups:
- PF-06463922 100 mg Single Dose (SD): PF-06463922 was administered following an overnight fast of at least 10 hours at approximately 0800 hours (plus or minus 2 hours) as 4 * 25 milligram (mg) tablets on Day 1 of Period 1. Investigator site personnel administered study medication with ambient temperature water to a total volume of approximately 240 milliliter (mL).
- Rifampin 600 Once a Day (QD) + PF-06463922 100 mg SD: Rifampin 600 mg once daily was administered 1 hour before or 2 hours after a meal from Day 1 to Day 9 of Period 2, except for rifampin dose on Day 8 of Period 2, which was administered simultaneously with PF-06463922. PF-06463922 100 mg (4 * 25 mg tablets) and rifampin were administered (rifampin followed by PF-06463922) following an overnight fast of at least 10 hours at approximately 0800 hours (plus or minus 2 hours).
Period: Period 1
Arm/Group | PF-06463922 100 mg Single Dose (SD) | Rifampin 600 Once a Day (QD) + PF-06463922 100 mg SD
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0
Period: Washout Period at Least 10 Days
Arm/Group | PF-06463922 100 mg Single Dose (SD) | Rifampin 600 Once a Day (QD) + PF-06463922 100 mg SD
Started | 12 | 0
Completed | 12 | 0
Not Completed | 0 | 0
Period: Period 2
Arm/Group | PF-06463922 100 mg Single Dose (SD) | Rifampin 600 Once a Day (QD) + PF-06463922 100 mg SD
Started | 0 | 12
Completed | 0 | 11
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study: All participants who received PF-06463922, rifampin and PF-06463922 in Period 1 and 2, respectively. A washout period of at least 10 days between the 2 single PF-06463922 dose was maintained.
Arm/Group | Entire Study
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.5 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Plasma AUCinf for PF-06463922 Given Alone and With Rifampin
Description: AUCinf is the plasma area under the plasma concentration-time profile from time 0 extrapolated to infinite time. The pharmacokinetics (PK) parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, 120 hours postdose on Day 1 after PF-06463922 100 mg administration in Period 1, and at the same time points on Day 8 after PF-06463922 100 mg with rifampin administration in Period 2.
Population: All participants who received PF-06463922, rifampin and PF-06463922 in Period 1 and 2, respectively. A washout period of at least 10 days between the 2 single PF-06463922 dose was maintained. Here, "Number of Participants analyzed" signifies number of participants evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram (ng)*hr/ millilitre (mL)
Groups:
- PF-06463922 100 mg: PF-06463922 was administered following an overnight fast of at least 10 hours at approximately 0800 hours (plus or minus 2 hours) as 4 * 25 milligram (mg) tablets on Day 1 of Period 1.
- Rifampin 600 mg + PF-06463922 100 mg: Rifampin 600 mg once daily was administered 1 hour before or 2 hours after a meal from Day 1 to Day 9 of Period 2, except for rifampin dose on Day 8 of Period 2, which was administered simultaneously with PF-06463922. PF-06463922 100 mg (4 * 25 mg table) and rifampin were administered (rifampin followed by PF-06463922) following an overnight fast of at least 10 hours at approximately 0800 hours (plus or minus 2 hours).
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 11
nanogram (ng)*hr/ millilitre (mL) | 8766 (19) | 1299 (30)
Statistical Analysis 1: Comparison: PF-06463922 100 mg vs Rifampin 600 mg + PF-06463922 100 mg; Mixed model was fitted to obtain ratio of geometric means of Rifampin 600 mg QD + PF-06463922 100 mg SD (test) to PF-06463922 100 mg SD (reference) and the results are presented as percentage. 90% CI was calculated on ratio of geometric means; Test type: Superiority or Other; Ratio of Geometric Mean = 14.74, 90% CI 2-sided [12.78 to 17.01]

2. Primary Outcome: Plasma Cmax for PF-06463922 Given Alone and With Rifampin
Description: Cmax is the maximum observed plasma concentration. PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: as for outcome 1
Population: All participants who received PF-06463922, rifampin and PF-06463922 in Period 1 and 2, respectively. A washout period of at least 10 days between the 2 single PF-06463922 dose was maintained.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 621.4 (26) | 148.4 (31)
Statistical Analysis 1: Comparison: PF-06463922 100 mg vs Rifampin 600 mg + PF-06463922 100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of Geometric Mean = 23.88, 90% CI 2-sided [21.58 to 26.43]

3. Secondary Outcome: Plasma AUClast for PF-06463922 Given Alone and With Rifampin
Description: AUClast is the plasma area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
ng•hr/mL | 8597 (19) | 1200 (32)
Statistical Analysis 1: Comparison: PF-06463922 100 mg vs Rifampin 600 mg + PF-06463922 100 mg; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; Ratio of Geometric Mean = 13.96, 90% CI 2-sided [12.09 to 16.12]

4. Secondary Outcome: Plasma Tmax for PF-06463922 Given Alone and With Rifampin
Description: Tmax is the time for maximum observed plasma concentration (Cmax). The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
hr | 1.50 [0.683 to 2.00] | 1.51 [1.00 to 4.00]

5. Secondary Outcome: Plasma t1/2 for PF-06463922 Given Alone and With Rifampin
Description: Terminal plasma half-life (t1/2) is the time measured for the plasma concentration of drug to decrease by one half. The PK parameter analysis population is defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 11
hr | 21.22 (4.12) | 10.16 (2.43)

6. Secondary Outcome: Plasma CL/F for PF-06463922 Given Alone and With Rifampin
Description: CL/F is the apparent oral clearance. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 11
L/hr | 11.39 (20) | 76.91 (30)

7. Secondary Outcome: Plasma Vz/F for PF-06463922 Given Alone and With Rifampin
Description: Vz/F is the apparent volume of distribution (only after single dose).The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: Predose, 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, 120 hours postdose on Day 1 after PF-06463922 100 mg administration in Period 1, and at the same time points on Day 8 after PF-06463922 100 mg administration with rifampin in Period 2.
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 11
liter | 342.6 (19) | 1095 (47)

8. Secondary Outcome: Plasma AUClast for PF-06895751 When PF-06463922 Given Alone and With Rifampin
Description: AUClast was the plasma area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period. PF-06895751 was the metabolite of PF-06463922.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 4105 (33) | 3169 (60)

9. Secondary Outcome: Plasma AUCinf for PF-06895751 When PF-06463922 Given Alone and With Rifampin
Description: AUCinf was the area under the plasma concentration-time profile from time 0 extrapolated to infinite time. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period. PF-06895751 was the metabolite of PF-06463922.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng•hr/mL
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 10 | 11
ng•hr/mL | 4453 (38) | 3291 (60)

10. Secondary Outcome: Plasma Tmax for PF-06895751 When PF-06463922 Given Alone and With Rifampin.
Description: Tmax was the time for maximum observed plasma concentration (Cmax). The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period. PF-06895751 was the metabolite of PF-06463922.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
hr | 30.1 [24.0 to 36.1] | 12.0 [6.00 to 36.1]

11. Secondary Outcome: Plasma t1/2 for PF-06895751 When PF-06463922 Given Alone and With Rifampin
Description: T1/2 was the terminal plasma half-life. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period. PF-06895751 was the metabolite of PF-06463922.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 10 | 11
hr | 29.14 (7.54) | 18.43 (4.10)

12. Secondary Outcome: Plasma Cmax for PF-06895751 When PF-06463922 Given Alone and With Rifampin
Description: Cmax was the maximum observed plasma concentration. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period. PF-06895751 was the metabolite of PF-06463922.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
ng/mL | 59.02 (29) | 76.45 (38)

13. Secondary Outcome: Plasma Molecular Weight Adjusted Metabolite to Parent (M/P) Ratio for Cmax (MRCmax) of PF-06463922 and Its Metabolite: When PF-06463922 Given Alone and With Rifampin
Description: Cmax was the maximum observed plasma concentration of PF-06463922 and PF-06895751 ( metabolite of PF-06463922). The molecular weight adjusted metabolite/parent ratio (PF-06895751/PF-06463922) for Cmax was presented. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
ratio | 0.2094 (29) | 1.136 (35)

14. Secondary Outcome: Plasma Molecular Weight Adjusted Metabolite to Parent (M/P) Ratio for AUClast (MRAUClast) of PF-06463922 and Its Metabolite: When PF-06463922 Given Alone and With Rifampin
Description: AUClast was the plasma area under the plasma concentration-time profile from time 0 to the time of the last quantifiable concentration of PF-06463922 and PF-06895751 ( metabolite of PF-06463922). The molecular weight adjusted metabolite/parent ratio (PF-06895751/PF-06463922) for AUClast was presented. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period. PF-06895751 was the metabolite of PF-06463922.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
ratio | 1.053 (24) | 5.831 (56)

15. Secondary Outcome: Plasma Molecular Weight Adjusted Metabolite to Parent (M/P) Ratio for AUCinf (MRAUCinf) of PF-06463922 and Its Metabolite: When PF-06463922 Given Alone and With Rifampin
Description: AUCinf was the plasma area under the plasma concentration-time profile from time 0 extrapolated to infinite time of PF-06463922 and PF-06895751 ( metabolite of PF-06463922). The molecular weight adjusted metabolite/parent ratio (PF-06895751/PF-06463922) for AUCinf was presented. The PK parameter analysis population was defined as all participants enrolled and treated who have at least 1 of the PF-06463922 PK parameters of primary interest in at least 1 treatment period.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 10 | 10
ratio | 1.166 (25) | 5.521 (56)

16. Other Pre Specified Outcome: Number of Participants With End of Study Abnormal Laboratory Findings Meeting the Criteria of Potentially Significant Clinical Concern
Description: The total number of participants with laboratory test abnormalities was assessed. Clinical laboratory tests included hematology, chemistry, urinalysis and some other tests (including follicle-simulating hormone[FSH], urine drug screening, hepatitis B surface antigen [HBsAg], hepatitis B core antibody [HBcAb], hepatitis C virus antibody [HCVAb] and human immunodeficiency virus [HIV]. Clinical significance was judged by the investigator.
Time Frame: Baseline to about 18 days after the first PF-06463922 dose
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Rifampin 600 mg QD: Rifampin 600 mg once daily was administered 1 hour before or 2 hours after a meal for 9 days, except for rifampin dose on Day 8, which was administered simultaneously with PF-06463922.
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg QD | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  No. of Participants Evaluable for Lab. Abnormality | 12 | 12 | 12
  No. With Lab. Abnormalities | 5 | 6 | 11

17. Other Pre Specified Outcome: Number of Participants With Physical Examination Findings Meeting the Criteria of Potentially Significant Clinical Concern
Description: A full physical examination included head, ears, eyes, nose, mouth, skin, heart and lung examinations, lymph nodes, gastrointestinal, musculoskeletal, and neurological systems. The limited or abbreviated physical examination focused on general appearance, the respiratory and cardiovascular systems, as well as towards participant reported symptoms. Clinical significance was judged by the investigator.
Time Frame: Baseline to about 18 days after the first PF-06463922 dose.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

18. Other Pre Specified Outcome: Number of Participants With Changes From Baseline and Absolute Values in Vital Signs Meeting the Criteria of Potentially Significant Clinical Concerns
Description: Criteria for potentially clinically important changes in vital signs were defined as: supine and standing systolic blood pressure (SBP) of less than (<90) millimeters of mercury (mm Hg) or change in supine and standing SBP more than or equal to (>=) 30 mm Hg; supine and standing diastolic blood pressure (DBP) of < 50 mm Hg or change in supine and standing DBP of >= 20 mm Hg; supine and standing pulse rate of < 40 or >120 beats per minute (bpm). Figure "99999" signifies data not measurable/applicable. Maximum Decrease is abbreviated as Max.Dec., and Maximum Increase is abbreviated as Max.Inc. n is the number of participants contributing to the parameter, not applicable is abbreviated as N/A.
Time Frame: Baseline to about 18 days after the first PF-06463922 dose.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
Participants
  Supine SBP (mmHg) <90 | 0 | 1
  Standing SBP (mmHg) <90: number analyzed (Participants) | 0 | 1
  Standing SBP (mmHg) <90 |  | 0
  Supine DBP (mmHg) <50 | 0 | 0
  Standing DBP (mmHg) <50: number analyzed (Participants) | 0 | 1
  Standing DBP (mmHg) <50 |  | 0
  Supine PR (BPM) >120 | 0 | 0
  Supine PR (BPM) <40 | 0 | 0
  Standing PR (BPM) >120: number analyzed (Participants) | 0 | 1
  Standing PR (BPM) >120 |  | 0
  Standing PR (BPM) <40: number analyzed (Participants) | 0 | 1
  Standing PR (BPM) <40 |  | 0
  Max.Dec. From Baseline in Supine SBP (mm Hg) >=30 | 0 | 0
  Max.Dec. From Baseline in Supine DBP (mm Hg) >=20 | 0 | 0
  Max.Inc. From Baseline in Supine SBP (mm Hg) >=30 | 0 | 1
  Max.Inc. From Baseline in Supine DBP (mm Hg) >=20 | 0 | 0

19. Other Pre Specified Outcome: Number of Participants With Electrocardiogram (ECG) Findings Meeting the Criteria of Potentially Significant Clinical Concerns
Description: PR interval was the interval between the start of the P wave and the start of the QRS complex, corresponding to the time between the onset of the atrial depolarization and onset of ventricular depolarization. Criteria for potentially clinically important changes (chg) in ECG were defined as: absolute values of PR interval >=200 to <220 msec, >=220 to <240 msec, >=240 to <260 msec and >=260 msec. Increase from baseline >=40, <60, >=60 and <80, >=80, and relative change from baseline >25%. The beginning of the Q wave to the end of the T wave corresponding to electrical systole (QT) interval corrected using the Fridericia formular (QTCF) of 450 to <480 msec, 480 to <500 msec and >=500 msec, or an increase of 30 to <60 msec of >=60 msec. Maximum is abbreviated as Max.
Time Frame: Baseline to about 18 days after the first PF-06463922 dose.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
Participants
  Maximum (Max) PR Interval (msec) 200-<220 | 0 | 0
  Max PR Interval (msec) 220-<240 | 0 | 0
  Max PR Interval (msec) 240-<260 | 0 | 0
  Max PR Interval (msec) >=260 | 0 | 0
  Max QT Interval (msec) >=500 | 0 | 1
  Max QTCF Interval (msec) 450-<480 | 0 | 1
  Max QTCF Interval (msec) 480-<500 | 0 | 0
  Max QTCF Interval (msec) >=500 | 0 | 0
  Max PR Interval Inc. From Baseline (msec) 40-<60 | 0 | 0
  Max PR Interval Inc. From Baseline (msec) 60-<80 | 0 | 0
  Max PR Interval Inc. From Baseline (msec) >=80 | 0 | 0
  Max PR Interval Inc.From Baseline(msec)PctChg>25% | 0 | 0
  Max QTCF Inc. From Baseline (msec) 30<=Chg<60 | 0 | 1
  Max QTCF Inc. From Baseline (msec) Chg>=60 | 0 | 0

20. Other Pre Specified Outcome: Number of Participants With Concomitant Treatments Meeting the Criteria of Potentially Significant Clinical Concerns
Description: Participants abstained from all concomitant treatments, except for the treatment of adverse events. Limited use of non-prescription medications that were not believed to affect participant safety or the overall results of the study might be permitted on a case by case basis following approval by the sponsor. All participants were questioned about concomitant treatment at each clinic visit. Treatments taken within 28 days before the first dose of study investigational product were documented as a prior treatment. Treatment taken after the first dose of study investigational product were documented as concomitant treatments. Females taking hormone replacement therapy might be eligible to participate in this study if they were willing to discontinue therapy at least 28 days prior to the first dose of study treatment and remained off hormonal therapy for duration of the study. Clinical significance was judged by the investigator.
Time Frame: Baseline to about 18 days after the first PF-06463922 dose.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12
Participants | 0 | 0

21. Other Pre Specified Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) (All Causalities and Treatment-Related)
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device; the event need not necessarily have a casual relationship with the treatment or usage. A serious adverse event (SAE) was any untoward medical occurrence at any dose that: 1) resulted in death; 2) was life threatening (immediate risk of death); 3) required inpatient hospitalization or prolongation of existing hospitalization; 4) resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); 5) resulted in congenital anomaly/birth defect. TEAE included both non-serious adverse events and serious adverse events.
Time Frame: Baseline to about 18 days after the first PF-06463922 dose.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg QD | Rifampin 600 mg + PF-06463922 100 mg
Number analyzed (Participants) | 12 | 12 | 12
Participants
  No. of Participants with AEs (all Causalities) | 1 | 5 | 12
  No. of Participants with SAEs (all Causalities) | 0 | 0 | 5
  Participants with Severe AEs (all Causalities) | 0 | 0 | 7
  Discontinued due to AEs (all Causality) | 0 | 0 | 12
  No. of Participants with AEs (Treatment Related) | 1 | 4 | 12
  No. of Participants with SAEs (Treatment Related) | 0 | 0 | 5
  Participants with Severe AEs (Treatment Related) | 0 | 0 | 7
  Discontinued due to AEs (Treatment Related) | 0 | 0 | 12

ADVERSE EVENTS:
Arm/Group | PF-06463922 100 mg | Rifampin 600 mg QD | Rifampin 600 mg + PF-06463922 100 mg
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 5/12
Other Adverse Events (participants affected / at risk) | 1/12 | 5/12 | 11/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06463922 100 mg (N=12) | Rifampin 600 mg QD (N=12) | Rifampin 600 mg + PF-06463922 100 mg (N=12)
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | PF-06463922 100 mg (N=12) | Rifampin 600 mg QD (N=12) | Rifampin 600 mg + PF-06463922 100 mg (N=12)
Dry eye (Eye disorders) | 0 | 1 | 1
Photophobia (Eye disorders) | 0 | 1 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 1
Defaecation urgency (Gastrointestinal disorders) | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 2
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 9
Retching (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3
Asthenia (General disorders) | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 1
Hangover (General disorders) | 0 | 0 | 1
Hunger (General disorders) | 0 | 0 | 1
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 0 | 7
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 2
Muscle twitching (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0 | 3
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
As all participants receiving co-administration of PF-06463922 (100 mg SD) with rifampin (600 mg QD) experienced drug-induced liver injury AEs, all 12 participants were discontinued from further rifampin treatment after 9 days but not 12 days.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No